CLINICAL TRIAL: NCT05682040
Title: Effect of Emergency Department Bedside Compression Ultrasonography on Door-to-Disposition Time in Patients Suspicious for Lower Extremity Deep Venous Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Christopher Nedzlek, Staff physician emergency department, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11243
Record Dates: First submitted 2022-12-14; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Lower Extremity Deep Vein Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Active (Other)
  Interventions: Diagnostic Test: Bedside Compression Ultrasonography

INTERVENTIONS:
Diagnostic Test: Bedside Compression Ultrasonography — Point of Care Ultrasound (Bedside Compression Ultrasonography) vs formal lower extremity Doppler

SUMMARY:
Comparing the disposition time of point of care ultrasound (POCUS) versus formal lower extremity doppler in emergency department patients.

ELIGIBILITY:
Inclusion Criteria: Emergency Department patients presenting for lower extremity swelling concerning Deep vein thrombosis.

-

Exclusion Criteria: n/a

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Time to disposition | 3 months
  We measured the time to disposition from the emergency department for point of care ultrasound (POCUS) vs formal lower extremity (LE) doppler in radiology department.

SECONDARY OUTCOMES:
Accuracy of POCUS vs formal LE doppler | 3 months
  We examined the accuracy of POCUS vs formal doppler in making the diagnosis of lower extremity deep vein thrombosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Wyandotte Hospital, Wyandotte, Michigan, United States

IPD SHARING:
Plan to Share IPD: No